CLINICAL TRIAL: NCT05115136
Title: The Use of Doxepin for Urticaria in the Emergency Department
Brief Title: Using Doxepin for Urticaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, David Andonian, Principal Investigator, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1576028
Record Dates: First submitted 2021-10-05; First posted 2021-11-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — Doxepin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Doxepin (Experimental): 25mg PO one time
  Interventions: Drug: Doxepin
- Diphenhydramine (Active Comparator): 50mg PO one time
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Doxepin — 25mg dose of Doxepin will be administered one time, by mouth
  Arms: Doxepin
Drug: Diphenhydramine — 50 mg dose of Diphenhydramine will be administered one time, by mouth
  Arms: Diphenhydramine

SUMMARY:
Isolated urticaria in the emergency department is widely treated by physicians with histamine blocking agents such as diphenhydramine, cetirizine, and cimetidine. Doxepin is a tricyclic antidepressant that has been shown to have much higher concentrations of histamine blocking activity and therefore may be useful in treating urticaria. The purpose of this study is to compare the effectiveness of using doxepin verses a traditional medication, diphenhydramine (Benadryl), in the treatment of isolated urticaria in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years of age
* Presenting to Upstate Adult Emergency Department at either the Downtown or Community campuses.
* Diagnosed with isolated/acute urticaria
* Requires treatment with antihistamines to alleviate symptoms

Exclusion Criteria:

* Pregnant women
* Prisoners
* Patients with altered mental status/have impaired decision-making capacity.
* Presenting with symptoms suggesting life threatening illness or anaphylaxis.
* Patients who have received any antihistamine (H1 antagonist) within the past 2 hours via any route of administration.
* Patients who have received an H2 antagonist within the past 2 hours.
* Patient received steroids by any route within the past 4 hours.
* Patient received epinephrine within the past 20 minutes.
* Patients currently taking concomitant p-glycoprotein inhibitors.
* Patients on any of the following CYP2D6 inhibitors: Bupropion, Fluoxetine, Paroxetine, Quinidine, Tipranavir.
* Patients with a history of serotonin syndrome.
* Patients currently taking another tricyclic antidepressant, selective serotonin reuptake inhibitor, and/or serotonin-norepinephrine reuptake inhibitor.
* Patients who have a condition where an antihistamine may be contraindicated.
* Patients with a contraindication to anticholinergic medications.
* History of adverse effects to tricyclic antidepressants or antihistamines.
* Patient who, based on their medical history or in the opinion of the clinician, have chronic urticaria, urticaria refractory to antihistamines, or dermatological disease that interferes with evaluation of a therapeutic response.
* Patients taking antileukotriene compounds (montelukast), calcineurin inhibitors (tacrolimus) or anti-serotonin agents (cyproheptadine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of urticaria | 1 hour after med administration, 2 hours after administration, and prior to discharge.
  Improvement of urticaria based on pruritis score. Scale is from 1-5, lower the score the better.
Improvement of urticaria | 1 hour after med administration, 2 hours after administration, and prior to discharge
  Improvement of urticaria based percent of body area affected. Scale being utilized is the % of body area chart.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No